CLINICAL TRIAL: NCT07346040
Title: Health Support Project for Persons With Disabilities
Acronym: JCHSP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Chair Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P0045968; P0045968 (Other Grant/Funding Number: The Hong Kong Jockey Club Charities Trust)
Record Dates: First submitted 2025-12-20; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Disabilities
Keywords: People with disabilities; Chronic diseases; Nutrition; Physical activity; Self-management
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Masking Description: No masking strategies will be included.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): We will use a waiting-list control group. People with disabilities in the control group will receive care as usual at study sites, be free to seek any health services during the study period, and be invited to join the HSP program for 24 weeks after the study ends
- Intervention group (Experimental): The intervention will last for 24 weeks.
  Interventions: Behavioral: Health Support Program

INTERVENTIONS:
Behavioral: Health Support Program — The Health Support Program (HSP) is a structured, multi-component intervention. The nutrition component will consist of one 45-minute [for those without intellectual disability (ID)] or 30-minute [for ID participants] group-based healthy eating education session per week, led by registered dietitians. The physical activity component will consist of three 30-minute sessions per week led by registered physiotherapists, together with the encouragement of community exercise and walk every day. Self-management of chronic conditions component will be implemented weekly in a 45-minute [for non-ID participants] or 30-minute [for ID participants] education session in a group format, which will be led by occupational therapists and nurses. To accommodate cognitive deficits in participants with ID and maximize their learning outcomes, additional support will be provided in terms of the structure (e.g., interactive format) of the intervention.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the health status of people with disabilities, to improve their health outcomes by providing support on nutrition, physical activity, and self-management of chronic conditions, and to strengthen sectors' capacity to deliver health management services and support for people with disabilities through a train-the-trainer program.

DETAILED DESCRIPTION:
In sheltered workshops (SWs) and integrated vocational rehabilitation services centers (IVRSCs) across Hong Kong, people with disabilities (PWDs) are provided with one-stop, integrated, and seamless vocational rehabilitation services in a specially designed environment. The aim is to help PWDs develop their social and economic potential to the fullest extent. Comorbid disorders - often overlooked when relevant sectors (e.g., non-government organizations) or healthcare professionals fail to look beyond disabilities - are likely to impose additional burdens on existing workload, resulting in adverse effect on their performance in areas such as productivity, health outcomes, personal well-being, and quality of life. Poor management of comorbid disorders may even lead to increased morbidity and mortality rates.

The Health Support Program (HSP) is a structured, multi-component intervention developed in close collaboration with a multidisciplinary research team of occupational therapists, physiotherapists, dietitians, and nurses from the Department of Rehabilitation Sciences and the Department of Food Science and Nutrition at The Hong Kong Polytechnic University. The program consists of three components: (1) nutrition, (2) physical activity, and (3) self-management of chronic conditions. The intervention is rooted in the Health Belief Model, and each component is developed based on international guidelines and current research findings. The HSP is tailored for PWDs with or without intellectual disabilities to improve health outcomes and is delivered with the assistance of the Digital Health Profile (DHP) System for the PWDs in the SWs and IVRSCs.

The DHP is a centralized database designed to record the health conditions of PWDs and optimize workflow management. Supported by an interactive dashboard and e-resources on health management, the core function of the DHP is to create health profiles for each PWDs, so that trained personnel from the SWs and IVRSCs can monitor and manage the health status of each PWDs more effectively and accurately. The DHP in all SWs and IVRSCs can together produce a comprehensive overview of the health conditions of PWDs in the community, which could facilitate and provide useful information for policy making.

Eligible PWDs in the SWs and IVRSCs who have at least one of the following physician-diagnosed chronic conditions: diabetes, hypertension, hyperlipidemia, cardiovascular disease, or obesity, will be recruited in a pragmatic, open-label, parallel-group, cluster-randomized clinical trial. The implementation of the HSP will be evaluated using the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) Framework.

ELIGIBILITY:
Inclusion Criteria:

* People with disabilities in sheltered workshops and integrated vocational rehabilitation services centers who had at least one of the following physician-diagnosed chronic conditions: diabetes, hypertension, hyperlipidaemia, cardiovascular disease, or obesity

Exclusion Criteria:

* Those with severe intellectual disabilities (IQ below 35) or at imminent risk of suicide

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Comprehensive health literacy | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Comprehensive health literacy will be measured as general knowledge of nutrition, physical exercise, and self-management of chronic diseases using a self-designed, closed-ended questionnaire. Responses will be scored as follows: 1 point for the correct answer, and 0 points for the incorrect answer or for the "Not sure" response. The dichotomized scores for each item in each area will be summed, with results ranging from 0 to 30 for knowledge of nutrition, 0 to15 for knowledge of physical activity, and 0 to 27 for knowledge of self-management of chronic diseases. For participants with intellectual disabilities, the number of items will be reduced. The results will range from 0 to 21 for knowledge of nutrition, 0 to15 for knowledge of physical activity, and 0 to 27 for knowledge of self-management of chronic diseases. Higher scores indicate better health literacy regarding nutrition, physical exercise, and self-management of chronic diseases, separately.

SECONDARY OUTCOMES:
Dietary intake | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Dietary intake will be captured via a self-designed, closed-ended questionnaire that asks individuals about the frequency of their consumption of 12 food items on a weekly basis. Participants will rate their weekly consumption of each food item on a 5-point Likert scale. On this scale, less healthy food items will be rated from daily consumption (0) to never consumption (4), while healthy food items will be rated in reverse, from daily consumption (4) to never consumption (0). In addition, there is 1 item, "Do you think your dietary habit is health", with responses is rating from "very unhealthy" (0) to "very health" (4). Total scores will range from 0 to 52, with higher scores indicating a healthier diet. For those with intellectual disabilities, the food items will be shorted to 8, with 6 less healthy food items and 2 healthy food items, resulting a total of score ranged from 0 to 32.
Achievement of physical activity goals | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Achievement of physical activity goals will be retrieved from each sheltered workshops and integrated vocational rehabilitation services centers if individuals meet the World Health Organization's recommendation of at least 150 minutes of moderate-intensity physical activity per week. The scoring system is dichotomous as: a "yes" response receives 1 point, and a "no" response receives 0 points.
Self-efficacy for physical activity | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Self-efficacy for physical activity will be assessed using the Chinese version of Self-Efficacy for Exercise (SEE) scale. The SEE evaluates individuals' perceived confidence in overcoming nine barriers to regular exercise: weather, boredom, pain, exercising alone, not pleasurable, too busy, feel tired, stress, depressed. For each situation, individuals rate their current confidence in exercising three times per week for 20 minutes each time using an 11-point Likert scale ranging from 0 (Not confident) to 10 (Very confident). The total score ranges from 0 to 90, with higher scores reflecting stronger levels of self-efficacy for exercise. This scale will not be used for participants with intellectual disabilities.
Body mass index (BMI) | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Body mass index (BMI) will be calculated as the weight in kilograms (kg; measured to the nearest 0.1 kg while wearing light clothing and stand erect, barefoot) divided by the squared height in meters (measured to the nearest 0.1 centimeters).
Blood pressure | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Blood pressure will be collected twice after a five-minute rest in a sitting position, with a five-minute rest in between. Readings will be taken on the right arm when possible; otherwise, readings will be taken on the left arm for those with conditions that preclude the use of the right arm, using electronic automated sphygmomanometers. The second reading will be used in all analyses, unless missing. According to the national guidelines, hypertension is defined as a systolic blood pressure of 140 mmHg or higher, a diastolic blood pressure of 90 mmHg or higher, or both.
Handgrip strength | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Handgrip strength will be measured three times in kilograms to the nearest 0.1 kg for each hand using a digital dynamometer, with a 60-second rest in between. Participants will be instructed to keep their elbow at a 90° angle flexion while either standing or sitting, with a neutral wrist position, and upper arm set vertically against the trunk. Participants will be required to squeeze the handle as hard as possible for three seconds. Handgrip strength will be considered as the maximum value of the three measurements for each hand.
Medication adherence | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Medication adherence will be measured with the Chinese version of the eight-item Morisky Medication Adherence Scale (MMAS-8). The scale includes seven dichotomous yes/no questions and one question answered on a five-point Likert scale. For Item 1 through 7, each "no" response is rated as 1, and each "yes" response is rated as 0, except for Item 5, where the "yes" response is rated as 1 and the "no" response is rated as 0. Item 8 contributes a score between 0 (All the time) and 1 (Never) in 0.25-point increments on a 5-point scale that assesses how often patients forget to take their medications. Item 8 will be adjusted for participants with intellectual disabilities as follows: "Do you have difficulty remembering to take all your medication(s)?" In the adjusted Item 8, the response of "difficulty" or "not sure" will be coded as 0, while "without difficulty" will be coded as 1. The total score is the sum of all MMAS-8 items and ranges between 0 and 8.
Mental well-being | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Mental well-being will be assessed using the Chinese version of the World Health Organization-Five Well-Being Index (WHO-5). The WHO-5 consists of five items, each of which is scored on a 6-point Likert scale with response options ranging from 0 (At no time) to 5 (All of the time). The WHO-5 raw score ranges from 0 to 25 and is conventionally multiplied by 4 to give a percentage score from 0, representing the worst imaginable well-being, to 100, corresponding to the best imaginable state of subjective well-being. For participants with intellectual disabilities, responses will be scored on a 3-point Likert scale: 0 (At no time), 1 (Sometimes), and 2 (All of the time) The total score is obtained by summing the scores of the five items and multiplying the raw score by 10, resulting in a percentage score ranging from 0 (worst well-being) to 100 (best well-being).
Health-related QoL | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Health-related quality of life will be evaluated via the Chinese version of the EuroQoL-5 Dimension-5 Level (EQ-5D-5L) instrument. The EQ-5D-5L descriptive system consists of the dimension of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, and each dimension includes five response categories of 1 (no problem), 2 (slight problems), 3 (moderate problems), 4 (severe problems), and 5 (extreme problems). A total of 3,125 (55) possible health states exists that are derived from the combination of each level of each dimension, with "11111" and "55555" representing the best and worst health states, respectively. The utility score of EQ-5D-5L will be derived using the established Hong Kong value set by weighting each respondent's self-report health status to a single preference-based health index (utility scores). A higher score in EQ-5D-5L will indicate better health-related quality of life.
Productivity levels | Baseline, 12-week mid-intervention, 24-week post-intervention, and 6-month follow-up
  Productivity levels improved after the launch of the Health Support Program. This improvement will be reflected in statistics from non-governmental organizations, particularly the total number of completed tasks by the people with disabilities in sheltered workshops and integrated vocational rehabilitation services centers.
Satisfaction levels | 12-week mid-intervention, 24-week post-intervention
  The satisfaction levels of participants will be rated on a 5-point Likert scale, ranging from"lowest satisfaction" (1) to "highest satisfaction" (5) for each component of the HSP intervention.

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication with no end date